CLINICAL TRIAL: NCT00901875
Title: An Open Multi-center Trial of Suboxone® (Buprenorphine/Naloxone) Treatment Among Opiate-Dependent Subjects
Brief Title: Multicentre Trial of Suboxone in Opiate-dependent Subjects in Taiwan
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Collaborators: Taipei City Psychiatric Center, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BU0808
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2010-01

CONDITIONS: Opiate Dependence
Keywords: Buprenorphine; Naloxone; Suboxone
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Naloxone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Suboxone, maximum 8mg (Experimental)
  Interventions: Drug: Buprenorphine + naloxone (Suboxone)
- Buprenorphine + naloxone (Experimental)
  Interventions: Drug: Buprenorphine + naloxone (Suboxone)
- Buprenorphine + naloxone (Suboxone) (Experimental)
  Interventions: Drug: Buprenorphine + naloxone (Suboxone)

INTERVENTIONS:
Drug: Buprenorphine + naloxone (Suboxone) — Sublingual tablets
  Other Names: Suboxone
Drug: Buprenorphine + naloxone (Suboxone)
  Other Names: Suboxone

SUMMARY:
To determine whether Suboxone can be effectively used to treat Taiwanese ethnic subjects with opiate dependence.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 20 years of age or older at screening visit.
* Subjects must meet DSM-IV/COWS1,2 criteria for opiate dependence. (COWS total score ≥5)
* Subjects must have a positive urine drug screen (dipstick test) for an opiate or morphine at study entry
* Subject is seeking treatment with the desire to discontinue opiate use as an initial goal but willing to consider and accept longer treatment if necessary.
* Subject is in good physical health or, if he/she has a medical condition needing ongoing treatment, must be in the care of a physician who is willing to take responsibility for such treatment and work with the study physician. Study physicians able to manage the subject for his/her general medical condition, may be assigned this role. These same conditions apply in case of subjects with psychiatric disorder(s) needing ongoing treatment.
* Subject is agreeable to and capable of signing informed consent form.
* Females of childbearing potential must have a negative pregnancy test and agree to use a double barrier method or condoms/diaphragm and spermicide contraceptive method during the study.

Exclusion Criteria:

* Women who are pregnant, lactating or breast feeding.
* Subjects have any acute medical condition that would make participation, in the opinion of the treating physician or the principal investigator, medically hazardous (e.g., acute hepatitis, unstable cardiovascular, liver or renal disease).
* Subjects have clinically significant liver disease.
* Subjects who have demonstrated a previous hypersensitivity to buprenorphine or naloxone.
* Subjects who are considered an immediate risk for suicide, are acutely psychotic, severely depressed, or in need of inpatient treatment.
* Subjects who are dependent on alcohol, benzodiazepines or other drugs of abuse (except tobacco) to the point of requiring immediate medical attention.
* Subjects received methadone treatment within the last 30 days since screening visit.
* Subjects have any pending legal action that could prohibit continued participation.
* Subjects have participated in other clinical studies within the past 30 days.
* Subjects who are expecting to leave the clinic geographic area prior to study completion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Retention in treatment | weekly up to 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Ku Lin, MD, Principal Investigator — Department of Psychiatry, Taipei City Psychiatric Center, Taipei, Taiwan.
Locations (8):
- Taiwan (8):
  - Jianan Mental Hospital, Rende, Tainan County
  - Taoyuan Mental Hospital, Taoyuan, Taoyuan County
  - Chang-Gung Memorial Hospital, Linkou Branch, Guishan
  - Chang-Gung Memorial Hospital, Keelung Branch, Keelung
  - China Medical University Hospital, Taichung
  - Taipei City Hospital - Song De Branch, Taipei
  - Taipei Veterans General Hospital, Taipei
  - BALI Psychiatric Center, Taipei